CLINICAL TRIAL: NCT03483155
Title: Compliance With The European Society Of Cardiology Prevention Guidelines In Patients at High Cardiovascular Disease Risk in Assiut University
Brief Title: Compliance With The European Society Of Cardiology Prevention Guidelines In Patients at High Cardiovascular Disease Risk
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noran Mohamed, Compliance With The European Society Of Cardiology Prevention Guidelines In Patients at High Cardiovascular Disease Risk in Assiut University, Assiut University
Other Study IDs: CESC
Record Dates: First submitted 2018-03-12; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Hypertension; Diabetes; Dyslipidemias
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with coronary or other atherosclerotic cardiovascular disease and those at high risk of developing cardiovascular disease have been defined as the highest clinical priorities for prevention

DETAILED DESCRIPTION:
Cardiovascular disease prevention programs are designed to reduce patients' morbidity and mortality.the European society of cardiology with other partner societies has engaged in a comprehensive programme of cardiovascular disease prevention in clinical practice aimed to improve practice of preventive cardiology by encouraging the development of national guidance on cardiovascular disease prevention

ELIGIBILITY:
Inclusion Criteria:

* Patients having signed an informed Consent Patients aged from 18 to 80 years old at the time of identification At least six and at most 24 months elapsed between the index event (the recruiting diagnostic or treatment criteria below) and the date of interview Patients meeting the recruiting diagnostic or treatment criteria: High CVD risk patients: patients free of CVD, who have been prescribed one or more of the following treatments: blood pressure and/or lipid-lowering and/or glucose lowering (diet and/or oral hypoglycaemic agents)

Exclusion Criteria:

* Patients living outside defined geographical area (Assiut Governorate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from hospital registries and general practice medical notes and will be interviewed between 6 months and 2 years after the date of recruiting event or procedure.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
the incidence of Cardiovascular disease | 18 months
  occurrence of any cardiovascular affection

CONTACTS AND LOCATIONS:
Overall Officials: Nouran Galal, Principal Investigator — AssiutUniversity

REFERENCES:
- [Background] EUROASPIRE. A European Society of Cardiology survey of secondary prevention of coronary heart disease: principal results. EUROASPIRE Study Group. European Action on Secondary Prevention through Intervention to Reduce Events. Eur Heart J. 1997 Oct;18(10):1569-82. doi: 10.1093/oxfordjournals.eurheartj.a015136. PMID 9347267
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren WM, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte Op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice; European Association for Cardiovascular Prevention and Rehabilitation. European Guidelines on cardiovascular disease prevention in clinical practice (version 2012): The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Atherosclerosis. 2012 Jul;223(1):1-68. doi: 10.1016/j.atherosclerosis.2012.05.007. Epub 2012 May 14. No abstract available. PMID 22698795
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] EUROASPIRE II Study Group. Lifestyle and risk factor management and use of drug therapies in coronary patients from 15 countries; principal results from EUROASPIRE II Euro Heart Survey Programme. Eur Heart J. 2001 Apr;22(7):554-72. doi: 10.1053/euhj.2001.2610. PMID 11259143
- [Background] EUROASPIRE I and II Group; European Action on Secondary Prevention by Intervention to Reduce Events. Clinical reality of coronary prevention guidelines: a comparison of EUROASPIRE I and II in nine countries. EUROASPIRE I and II Group. European Action on Secondary Prevention by Intervention to Reduce Events. Lancet. 2001 Mar 31;357(9261):995-1001. doi: 10.1016/s0140-6736(00)04235-5. PMID 11293642
- [Background] De Sutter J, De Bacquer D, Kotseva K, Sans S, Pyorala K, Wood D, De Backer G; EUROpean Action on Secondary Prevention through Intervention to Reduce Events II study group. Screening of family members of patients with premature coronary heart disease; results from the EUROASPIRE II family survey. Eur Heart J. 2003 Feb;24(3):249-57. doi: 10.1016/s0195-668x(02)00386-x. PMID 12590902
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. EUROASPIRE III: a survey on the lifestyle, risk factors and use of cardioprotective drug therapies in coronary patients from 22 European countries. Eur J Cardiovasc Prev Rehabil. 2009 Apr;16(2):121-37. doi: 10.1097/HJR.0b013e3283294b1d. PMID 19287307
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Reiner Z, Keil U; EUROASPIRE Study Group. EUROASPIRE III. Management of cardiovascular risk factors in asymptomatic high-risk patients in general practice: cross-sectional survey in 12 European countries. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):530-40. doi: 10.1097/HJR.0b013e3283383f30. PMID 20577089
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. Lancet. 2009 Mar 14;373(9667):929-40. doi: 10.1016/S0140-6736(09)60330-5. PMID 19286092
- [Background] Kotseva K, Ryden L, De Backer G, De Bacquer D, Wood D. EURObservational research programme: EUROASPIRE. Eur Heart J. 2015 Apr 21;36(16):950-1. doi: 10.1093/eurheartj/ehv047. No abstract available. PMID 25899410
- [Background] Gyberg V, De Bacquer D, Kotseva K, De Backer G, Schnell O, Sundvall J, Tuomilehto J, Wood D, Ryden L; EUROASPIRE IV Investigators. Screening for dysglycaemia in patients with coronary artery disease as reflected by fasting glucose, oral glucose tolerance test, and HbA1c: a report from EUROASPIRE IV--a survey from the European Society of Cardiology. Eur Heart J. 2015 May 14;36(19):1171-7. doi: 10.1093/eurheartj/ehv008. Epub 2015 Feb 9. PMID 25670820
- [Background] Gyberg V, De Bacquer D, De Backer G, Jennings C, Kotseva K, Mellbin L, Schnell O, Tuomilehto J, Wood D, Ryden L, Amouyel P, Bruthans J, Conde AC, Cifkova R, Deckers JW, De Sutter J, Dilic M, Dolzhenko M, Erglis A, Fras Z, Gaita D, Gotcheva N, Goudevenos J, Heuschmann P, Laucevicius A, Lehto S, Lovic D, Milicic D, Moore D, Nicolaides E, Oganov R, Pajak A, Pogosova N, Reiner Z, Stagmo M, Stork S, Tokgozoglu L, Vulic D; EUROASPIRE Investigators. Patients with coronary artery disease and diabetes need improved management: a report from the EUROASPIRE IV survey: a registry from the EuroObservational Research Programme of the European Society of Cardiology. Cardiovasc Diabetol. 2015 Oct 1;14:133. doi: 10.1186/s12933-015-0296-y. PMID 26427624
- [Background] Syntax score calculator. syntax working group. 5-19-2009. Ref Type: Electronic Citation